CLINICAL TRIAL: NCT02419105
Title: Effects of Transdermal Testosterone and/or Monthly Vitamin D on Fall Risk in Pre--frail Hypogonadal Seniors. Double Blind, 2x2 Factorial, Randomized Placebo--Controlled Clinical Trial
Brief Title: Effects of Transdermal Testosterone and/or Monthly Vitamin D on Fall Risk in Pre--frail Hypogonadal Seniors
Acronym: T&D
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Delayed recruitment mainly due to a screening to inclusion rate much lower than expected. Due to the delayed recruitment IMP reached the end of its shelf life.
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Besins Healthcare (funding: investigator-initiated and independent grant) (Unknown); Dr. Wild & Co. (funding: investigator-initiated and independent grant) (Unknown); Cantonal Hospital of St. Gallen (Other); Tufts University Jean Mayer USDA Human Nutrition Research Center on Aging (Other); Centre on Ageing and Mobility (Dr. Andreas Egli) (Unknown); University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T&D Study; 32003B_135192 (Other Grant/Funding Number: Swiss National Science Foundation); SNCTP: 000001224 (Registry Identifier: Swiss Clinical Trials Portal); KEK-ZH-2014-0436 (Other: Cantonal Ethics Committee Zurich, Switzerland); 2105DR3024 (Other: Swiss Agency for Therapeutic Products (Swissmedic))
Record Dates: First submitted 2015-03-30; First posted 2015-04-17 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Hypogonadism; Pre-frail Seniors
Keywords: Falls; hypogonadal men; Seniors; Testosterone; Colecalciferol
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Testosterone + Vitamin D (Active Comparator): Testosterone, transdermal gel, 75 mg, once per day, for 12 months AND Colecalciferol, oral drink solution, 24000 IU, once per month, for 12 months
  Interventions: Drug: Testosterone; Drug: Colecalciferol
- Testosterone + Placebo (Active Comparator): Testosterone, transdermal gel, 75 mg, once per day, for 12 months AND Placebo: Colecalciferol, oral drink solution, 0 IU, once per month, for 12 months
  Interventions: Drug: Testosterone; Drug: Placebo drink solution
- Placebo + Vitamin D (Active Comparator): Placebo: Testosterone, transdermal gel, 0 mg, once per day, for 12 months AND Colecalciferol, oral drink solution, 24000 IU, once per month, for 12 months
  Interventions: Drug: Colecalciferol; Drug: Placebo transdermal gel
- Control (Placebo Comparator): Placebo: Testosterone, transdermal gel, 0 mg, once per day, for 12 months AND Placebo: Colecalciferol, oral drink solution, 0 IU, once per month, for 12 months
  Interventions: Drug: Placebo drink solution; Drug: Placebo transdermal gel

INTERVENTIONS:
Drug: Testosterone — transdermal gel, 75 mg daily
  Other Names: ATC code: G03BA03
  Arms: Testosterone + Placebo; Testosterone + Vitamin D
Drug: Colecalciferol — drink solution, 24000 IU once per month
  Other Names: Vitamin D3, CAS No: 67-97-0, ATC code: A11CC05
  Arms: Placebo + Vitamin D; Testosterone + Vitamin D
Drug: Placebo drink solution — drink solution, 0 IU Colecalciferol once per month
  Arms: Control; Testosterone + Placebo
Drug: Placebo transdermal gel — transdermal gel, 0 mg testosterone daily
  Arms: Control; Placebo + Vitamin D

SUMMARY:
The overall purpose of this study is to test the individual and combined effect of transdermal testosterone and/or Vitamin D in reducing fall risk and improve function in pre-frail hypogonadal senior men.

DETAILED DESCRIPTION:
Background:

One of the challenges of demographic change is the enormous personal and economic burden of falls and their consequences in the senior population. Thirty percent of adults 65 years or older and 40 - 50% of those age 80 years or older fall once per year. Serious injuries occur in 10 - 15% of falls, resulting in fractures in 5% and a hip fracture in 1-2% of cases. As an independent determinant of functional decline, falls lead to 40% of all nursing home admissions.

Several studies have estimated the prevalence of low testosterone levels (hypogonadism) in older men to be about 20% at age 60. This proportion increased in the Baltimore Longitudinal Study of Aging with each decade (30% at age 70 and 50% at age 80). Low testosterone levels are associated with decreased strength, impaired physical performance, and an increased risk of falls, and, thus, low testosterone may contribute to the frailty syndrome in older men. Current studies have focused on healthy, community dwelling men with a high level of function. Our trial aims to enrol pre-frail senior men at risk of losing their autonomy. Further, in this population and also relevant for muscle health and falling is the high prevalence of vitamin D deficiency.

Dose Rationale:

The investigators chose 75 mg testosterone/day as the minimally sufficient dose to shift over 90% of participants to total testosterone levels of at least 16.86 nmol/l (lower end of the third quartile in the pilot trial where fall reduction was significant -- Bischoff-Ferrari et al.; Osteoporosis International 2008). Additionally, this dose has been chosen for its cardiovascular safety as summarized in a 2013 review.

The investigators chose 24000 IU/month of vitamin D (equivalent to 800 IU vitamin D per day) as the current recommended dose for vitamin D and its evidence for fall reduction. To allow for the standard of care and given that 50% of participants will not be randomized to vitamin D supplementation - all participants are allowed to take 800 IU vitamin D per day in addition to the study medication.

Randomization:

Participants will be randomized at the baseline clinical visit using a computer-based randomization procedure. Willing and eligible participants will be randomized to one of the four treatment groups stratified by age (2 groups: 75 - 79 and 80+). Within each stratum, treatment assignments will be generated in blocks of 8 individuals, with 2 individuals in each of the 4 treatment groups.

Blinding:

Study medications will be labelled with a unique randomization code at the respective companies. The codes will be inaccessible until the data set is frozen and the study is unblinded. All study packages will look identical, except for the randomization codes on the labels.

Follow-up:

Follow-up is 12 months with 3 clinical (Baseline, 6 and 12 months) and 4 (2, 4, 8 and 10 months) phone call visits.

Determination of Sample Size:

The sample size of 168 senior participants was chosen to have sufficient power for the primary endpoint (odds of falling) and the effect of testosterone treatment. Under these assumptions and assuming an additive effect of the 2 interventions (testosterone and vitamin D), as expected from the investigators pilot study, they have 89% power for the primary endpoint "number of participants sustaining at least 1 fall". This computation assumes that the difference in proportions of fallers is -0.24 (specifically, 0.38 versus 0.62 - based on the investigators pilot study). If 17% of participants would contribute no data (total n = 140), the investigators would still have 82% power to detect this difference.

Rate of falls: under the same assumptions, and with the proposed sample size of 84 and 84 for the two groups, the study will have power of at least 90.6% to yield a statistically significant result for the rate of falls. This computation assumes that the mean difference in rate of falls is -1.0 (corresponding to means of 0.9 versus 1.9) and the common within-group standard deviation is 2.0 (based on standard deviation estimates of 2.2 and 1.7).

Planned Analyses:

Primary analysis will be conducted according to the intention to treat (ITT) principle. Every study participant who was randomized and received the study treatment package at baseline clinical visit will be a part of the primary analysis population. In addition to the primary ITT analyses, the same data will be analyzed in participants who demonstrated acceptable adherence to the study protocol. The per protocol analyses will be treated as sensitivity analyses. The per protocol analysis population will include the participants who: Attended at least 1 out of the 2 follow-up clinical visits; Participated in at least 2 of the 4 follow-up phone calls; Took at least 80% of the study medication(s) as confirmed by count of used bottles for drinking solution and count and weight of used transdermal gel containers; did not take additional vitamin D and calcium supplements in doses exceeding those stipulated by the exclusion criteria.

All assessments of treatment effects in the efficacy analyses will be based on the intent-to-treat principle. All endpoint variables will be summarized by treatment group. N, Mean, Standard Deviation, Minimum and Maximum will summarize continuous endpoint variables and Number and Percentage will summarize categorical endpoint variables. All endpoints will be tested at the 2-sided at 5% significance level (α = 0.05, 2-sided). Two types of models will be run for each analysis. Minimally adjusted models will include age, body mass index, and baseline serum levels of total testosterone and 25-hydroxyvitamin D; fully adjusted models in addition to the parameters included in the minimally adjusted models will also include number of comorbidities, cognitive function, and additional potential confounders if baseline analysis justifies their inclusion. Each of the models will initially check for possible interaction between the study treatments. If no such interaction in found, the interaction term will be dropped and the simplified models will be used to estimate separate effects of the study treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Men with documented total testosterone levels < 11.30 nmol/l
2. Able to come to the study centre (Community-dwelling or institutionalized)
3. Age 65+ years
4. At a higher risk for falling
5. Body mass index > 18.0 and < 35.0 kg/m2
6. Understands German in reading and writing plus able to read, understand, and complete questionnaires and tests.
7. Willingness to limit additional vitamin D3 intake to a maximum of 800 IU per day
8. Willingness to limit calcium supplement intake to 500 mg/day
9. Willingness to stop active vitamin D metabolites
10. Willingness to forgo any additional use/application of testosterone products for the duration of the trial.
11. Participant understands the study procedures, alternative treatments available and risks involved with the study and voluntarily agrees to participate by giving a written informed consent.
12. Participant meets the routine clinical laboratory safety screening tests performed at screening visit.
13. Participant is able and willing to perform all study tests, attend all required office visits, and provide blood and urine samples.
14. Participant is able to apply the testosterone/placebo gel and is able to drink the vitamin D/placebo solution.
15. Participant is mentally competent (judicious) defined by having score > 24 on the Folstein's mini mental state examination (MMSE) at the screening visit.

Exclusion Criteria:

1. Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product
2. Treatment with vitamin K-antagonists, insulin, adrenocorticotropic hormone (ACTH), corticosteroid (>5mg/d)
3. Elevated (≥ 4.0 ng/ml) prostate-specific antigen levels (at screening) and/or palpable signs of prostate cancer
4. Palpable signs of breast-cancer
5. Haemoglobin ≤ 100 g/l
6. Haematocrit ≥ 0.50 L/L
7. Liver function values (alanine aminotransferase, aspartate aminotransferase, Gamma-glutamyl transferase, alkaline phosphatase) more than 3 times the upper limit of normal.
8. Consumption of >800 IU vitamin D on any day in the 6 months prior to enrolment. Provision: a person can be enrolled as soon as the mean intake in the last 6 months and since the last dose is ≤ 800 IU.
9. Elevated serum calcium ≥ 2.60 mmol/l (adjusted for albumin )
10. Estimated (Cockcroft and Gault formula ) creatinine clearance ≤ 30 ml/min
11. Severe visual or hearing impairment
12. History of cancer < 5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer
13. Myocardial infarction in the last 3 months, unstable angina pectoris and/or exertional dyspnoea >=NYHA III
14. Treatment worthy but untreated sleep apnoea or chronic (obstructive) pulmonary disease, epilepsy
15. Significant end-stage disease, i.e. genitourinary, cardiovascular, hepatic, renal, endocrine, hematologic, psychiatric, or pulmonary disease, which, in the opinion of the investigator, may pose a high risk to the patient or impair the patient's ability to complete the trial or confound the results
16. Uncontrolled hypertension (blood pressure mm Hg ≥ 180 systolic or ≥ 110 diastolic)
17. Alcohol abuse or alcoholic disease
18. Participation in another interventional research trial within the last 6 months prior to screening
19. Severe gait impairment, e.g. due to Parkinson's disease or hemiplegia
20. Previous enrolment into the current study
21. Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-09; Primary Completion 2020-05 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Number of fallers | 12 months
  The participant will fill in a falls diary.
Rate of falls | 12 months
  The participant will fill in a falls diary.

SECONDARY OUTCOMES:
Appendicular lean skeletal muscle mass (aLSM) | 12 months
  measured by dual energy X-ray absorptiometry (aLSM is defined as of skeletal muscles in upper and lower extremities)
Lower extremity function | 12 months
  assessed with the Short Physical Performance Battery (SPPB)
Reaction time | 12 months
  assessed by repeated sit-to-stand test (part of the SPPB)
Gait Speed | 12 months
  assessed by 4 meter walk test (part of the SPPB)
Quality of life | 12 months
  assessed by EuroQol (EQ5D-3L)

OTHER OUTCOMES:
Cognitive function | 12 months
  assessed by the Montreal Cognitive Assessment (MoCA) test
Body composition | 12 months
  measured by dual energy X-ray absorptiometry
Hip bone density | 12 months
  measured by dual energy X-ray absorptiometry
Incidence of sarcopenia | 12 months
  Since there is no consensus on a universally accepted definition of sarcopenia to date, all previously used and newly proposed composite definitions of sarcopenia based on lean mass and the SPPB, its components and/or grip strength, will be considered.
Bone quality (bone micro-architecture and bone strength) | 12 months
  measured by high-resolution peripheral quantitative computed tomography (XtremeCT)
serum concentrations of 25(OH)D | 12 months
  Adherence, Laboratory measures at the Institute of Clinical Chemistry at the University Hospital Zürich
free and bioavailable testosterone (serum concentration of total testosterone, sex hormone binding globulin, albumin) | 12 months
  Adherence, Laboratory measures at the Institute of Clinical Chemistry at the University Hospital Zürich, total testosterone will be measured, free and bioavailable testosterone will be calculated
haemoglobin, haematocrit, prostate-specific antigen, calcium, creatinine, alanine aminotransferase, aspartate aminotransferase, Gamma-glutamyl transferase, alkaline phosphatase | 12 months
  Laboratory measures at the laboratory of the City Hospital Waid, Zürich
Incidence of cardiovascular adverse events | 12 months
  "cardiovascular event" defined as: myocardial infarction, stroke, revascularization procedure of coronary artery bypass graft and percutaneous coronary intervention, incident congestive heart disease (heart insufficiency), cardiovascular mortality

CONTACTS AND LOCATIONS:
Overall Officials: Heike A Bischoff-Ferrari, MD, DrPH, Principal Investigator — University of Zurich
Locations (1):
- Dept. of Geriatrics and Aging Research, University of Zurich / Geriatric Clinic University Hospital Zurich, Zurich, Canton of Zurich, Switzerland